CLINICAL TRIAL: NCT00580385
Title: Chemotherapy Resistance in Osteogenic Sarcoma and Other Solid Tumors
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Hospital for Special Surgery, New York (Other); Weill Medical College of Cornell University (Other); Columbia University (Other); Rockefeller University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 97-094
Record Dates: First submitted 2007-12-20; First posted 2007-12-24 (Estimated); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Osteosarcoma
Keywords: BONE
MeSH Terms: conditions — Osteosarcoma | interventions — Tissue and Organ Procurement

ARMS (1):
- 1 (Experimental)
  Interventions: Other: Tissue Procurement

INTERVENTIONS:
Other: Tissue Procurement — MTX polyglutamylation, MTX transport, XTT cytotoxicity assays, Quantitative RT-PCR, Southern blotting, Mutation detection, and Western blotting

SUMMARY:
The purpose of this study is to investigate tumors in the laboratory to determine how and why they respond, or fail to respond to different drug therapies. This study will also investigate why high pressure develops within tumors and how this affects how well drugs work. We will also take blood samples before and/or after your procedure to measure biochemical factors that may help us predict the behavior of osteogenic sarcoma and other solid tumors.

DETAILED DESCRIPTION:
When tumor tissue known or presumed to be a primary or secondary bone cancer or solid tumor with known elevated intra-tumoral pressure such as retinoblastoma is being removed or has been removed for diagnostic or therapeutic reasons a small sample of it will be obtained for this study. The tumor samples will be used to study in vitro, determinants of chemotherapy resistance and oncogenesis. These determinants will be correlated with histologic response to preoperative chemotherapy and clinical outcome (event free survival). In addition, blood samples (20ml) may be obtained before or after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* All patients with a presumed or known diagnosis of a primary or secondary bone cancer or other solid tumor who are having or have had a biopsy or surgery to remove tumor for diagnostic or therapeutic reasons. No tumors will be obtained solely for research purposes.
* All adult patients (> or = to 18 yrs.) will have given written informed consent.
* All minor patients (<18 yrs.) will have given assent to the best of their ability to understand, and their parent or guardian will have given written informed consent

Exclusion Criteria:

* N/A

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 763 (Actual)
Dates: Start 1997-08; Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
To test tumor samples obtained from patients with primary or secondary bone cancer for mechanisms of acquired and intrinsic resistance to methotrexate and to relate these findings to histologic response to preoperative chemotherapy and outcome. | 2 years

SECONDARY OUTCOMES:
To attempt to grow these tumor cells in short term culture to test the sensitivity of these cells to chemotherapeutic agents and to correlate cytotoxicity with biochemical and molecular studies. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: John Healey, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org